CLINICAL TRIAL: NCT02611206
Title: Repetitive Transcranial Magnetic Stimulation for Adolescent Depression: Efficacy, Predictive Biomarkers, and Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSYCH-2016-18311
Record Dates: First submitted 2015-10-12; First posted 2015-11-20 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Treatment Resistant Depression
Keywords: rTMS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Period 1: 80% of MT (Experimental): All participants who qualify will undergo 6 weeks of open-label rTMS with a stimulation intensity of 80% of MT
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS): intensity 80% MT
- Period 2: 100% of MT (Experimental): All participants who qualify will undergo 6 weeks of open-label rTMS with a stimulation intensity of 100% of MT
  Interventions: Device: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Stimulation intesity: 100% of MT
- Period 3: 120% of MT (Experimental): All participants who qualify will undergo 6 weeks of open-label rTMS with a stimulation intensity of 120% of MT
  Interventions: Device: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Stimulation intesity: 120% of MT

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS): intensity 80% MT — rTMS applies a pulsatile magnetic field to the scalp which painlessly induces electrical currents to the brain. Typically, rTMS is applied to the dorsolateral prefrontal cortex (DLPFC), a brain region that is hypoactive in depression. Whereas standard rTMS stimulates superficial (1cm depth) cortical areas, recent advances in rTMS coil technology support stimulation of deeper (5 cm depth) limbic structures that are also relevant to depression.
  Other Name: Brainsway rTMS
  Other Names: Brainsway rTMS
  Arms: Period 1: 80% of MT
Device: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Stimulation intesity: 100% of MT — rTMS applies a pulsatile magnetic field to the scalp which painlessly induces electrical currents to the brain. Typically, rTMS is applied to the dorsolateral prefrontal cortex (DLPFC), a brain region that is hypoactive in depression. Whereas standard rTMS stimulates superficial (1cm depth) cortical areas, recent advances in rTMS coil technology support stimulation of deeper (5 cm depth) limbic structures that are also relevant to depression.
  Other Name: Brainsway rTMS
  Arms: Period 2: 100% of MT
Device: Device: Active Repetitive Transcranial Magnetic Stimulation (rTMS); Stimulation intesity: 120% of MT — rTMS applies a pulsatile magnetic field to the scalp which painlessly induces electrical currents to the brain. Typically, rTMS is applied to the dorsolateral prefrontal cortex (DLPFC), a brain region that is hypoactive in depression. Whereas standard rTMS stimulates superficial (1cm depth) cortical areas, recent advances in rTMS coil technology support stimulation of deeper (5 cm depth) limbic structures that are also relevant to depression.
  Other Name: Brainsway rTMS
  Arms: Period 3: 120% of MT

SUMMARY:
This study will be an open-label 6-week (30 session) trial of active repetitive transcranial magnetic stimulation (rTMS) using a fixed frequency (10 Hz) but varying stimulation intensities using a 3+3 study design for safety and tolerability amongst adolescents. This means that we will only enroll 3 participants at a time and give them rTMS at the stimulation intensity energy of 80% of motor threshold (MT). If all three participants complete the 6 weeks of treatment with no major safety events (i.e. seizure), we will increase the energy for the next 3 participants by 20%. If 1 of the 3 participants has a major safety event, we will enroll 3 more patients at the SAME energy. We will proceed in this manner, increasing by 20% after 3 subjects safely complete treatment at that energy, to a maximum energy of 120% of motor threshold. If 2 participants in each intensity level cohort experience a major safety event, we will discontinue running subjects at that energy level. If this happens at our initial energy level of 80% of MT, we will stop the study. If we reach 2 events in any of the higher energy cohorts, we will return to the previous energy level and complete the remainder of the subjects at that energy level.

DETAILED DESCRIPTION:
Adolescents with Treatment Resistant Depression (TRD) (n=30) will be recruited from the inpatient and outpatient adolescent mental health clinical services at UMN and surrounding area.

Adolescents and parents will undergo the consent process and initial clinical evaluation. This initial evaluation will be done using the Kiddie Schedule of Affective Disorders and Schizophrenia (K-SADS-PL 2009) and the Children's Depression Rating Scale-Revised (CDRS-R). Participants and their families will also be asked to complete the Antidepressant Treatment Report (ATR), Beck Depression Inventory (BDI-II), Columbia Suicide Severity Rating Scale (C-SSRS), Inventory of Depression and Anxiety Symptoms (IDAS), Temporal Experience of Pleasure Scale (TEPS), Snaith-Hamilton Pleasure Scale (SHAPS), Young Mania Rating Scale (YMRS), Edinburgh Handedness Scale, the Weschler Abbreviated Scale of Intelligence (WASI) and the Tanner Pubertal Staging Questionnaire. Participants will also be asked to complete the NIH Toolbox, Children's Auditory Verbal Learning Test (CAVLT), and the Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test.

Adolescents with TRD who fit inclusion/exclusion criteria (presence of major depression with CDRS-R raw score > 40; a history of at least one failed treatment trial with an antidepressant [as defined by the Antidepressant Treatment Report]; no history of seizure disorder; no presence of MRI contraindications [e.g. claustrophobia or metallic implants]) will be scheduled for:

A. A baseline MRI (described below)

B. 6 weeks of the series of rTMS visits described below

C. A post-treatment MRI

D. A post-treatment clinical assessment (blinded to treatment assignment)

E. 6 monthly follow up visits

In the first rTMS visit, the study physician will fit the cap, determine the ideal location for stimulation, and measure MT and MEPa. Adolescents will receive 6 weeks of rTMS, 20 minutes/day, 5 days/week administered by a trained technician. Active treatment will be 43 trains of 10 Hz, stimulation intensity will vary as described above, inter-train interval 20 seconds, 1680 pulses/session. A member of research staff will meet weekly with patients to complete the CDRS-R, monitor treatment tolerance using the Side Effects Form for Children and Adolescents, and measure the MT and MEPa. Adolescents will also complete the BDI-II, C-SSRS-SLV, IDAS, TEPS, YMRS, and SHAPS weekly. At week four, the participants will be asked to repeat the NIH Toolbox, Children's Auditory Verbal Learning Test (CAVLT), and the Delis-Kaplan Executive Function System (D-KEFS) Trail Making Test.

Scanning will take place at the Center for Magnetic Resonance Research on a 3T Siemens Prisma scanner at baseline (after the clinical assessment, before the first treatment) and after the last rTMS treatment. Participants will complete MRI safety forms and provide a urine sample to rule out substance use (all participants) and pregnancy (females only). A high-resolution T1 image will be collected (voxel size=1mm isotropic; TR=2530ms; TE=3.65ms, T1=1100ms, flip angle=7°, 5 minutes). Functional data will be acquired using the Human Connectome Project (HCP)38 multiband echo planar imaging sequence (whole brain T2*-weighted functional volumes, 72 contiguous slices; TR=720ms; TE=34.2ms; flip angle=55o, FOV=212mm; voxel size=2mm isotropic; matrix=106x106; multiband factor=8; 12 minutes) during rest with eyes open while viewing a fixation cross.

Participants will be asked to complete a task fMRI in which they are presented with a series of visual stimuli, (human faces of varying emotion expressions with positive, negative or neutral words printed over the faces). During the task, participants will be asked to decide whether the words printed over the faces are positive or negative regardless of the emotion of the face shown. Each subject will complete four distinct blocks of the task.

After the completion of rTMS sessions, all participants will undergo a final assessment during which they will be asked to meet with evaluators again to complete the CDRS-R. They will also be asked to complete the BDI-II, C-SSRS, TEPS, SHAPS, IDAS and NIH Toolbox.

After the completion of all rTMS sessions, participants will be asked to return to see researchers every month for 6 months to assess length of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD)
* A CDRS-R score of >40
* Experiencing a current MDD episode with a duration of ≥ 4 weeks and ≤3 years
* Resistance to treatment, defined by failure to respond adequately to at least one antidepressant treatment, defined by ATR level 1-4 in current episode
* Both child and parent/guardian are English speaking
* Female participants who are sexually active during the course of the study must use a form of birth control for the duration of the study

Exclusion Criteria:

* Any subject with a clinically defined neurological disorder or insult including, but not limited to, a condition likely to increase the risk of seizure; such as, space occupying brain lesion; any history of seizure; history of cerebrovascular accident; transient ischemic attack within two years; cerebral aneurysm; dementia; brain surgery; history or stroke or family history of epilepsy
* Any subject with an increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure or history of significant head trauma with loss of consciousness for ≥ 5 minutes
* Positive responses to any question on the Transcranial Magnetic Stimulation Adult Safety Screening Questionnaire (TASS)
* Subjects with cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute unstable cardiac diseases
* Subjects with conductive, ferromagnetic, or other magnetic-sensitive metals implanted in the head within 30 cm of the treatment coil excluding the mouth that cannot safely be removed should be excluded. Examples include cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes
* Subjects with active or inactive implants (including device leads), including deep brain stimulators, cochlear implants, and vagus nerve stimulators
* Inability to locate and quantify a motor threshold as defined in the protocol
* History of treatment with ECT or TMS therapy for any disorders
* Participation in any investigational drug trial within 4 weeks of the baseline visit
* Pregnancy
* IQ < 80
* Clinically significant laboratory abnormality or medical condition, that in the opinion of the investigator would hinder the subject in completing the procedures required by the study
* Suicide attempt within the previous 6 months that required medical treatment or ≥2 attempts in the past 12 months, or has a clear plan for suicide and states that s/he cannot guarantee that s/he will inform a family member or call his/her psychiatrist or the investigator if the impulse to implement the plan becomes substantial during the study; or, in the investigator's opinion, is likely to attempt suicide within the next 6 months
* Unstable psychotherapy (therapy must be for at least 3 months prior to entry into the study, with no anticipation of change in the frequency or treatment focus of the therapeutic sessions over the duration of the study)
* A diagnosis of substance use disorder, Schizophrenia, Bipolar Disorder, or Autism
* Refusal to cooperate with study procedures
* Recent change in dose of antidepressant medication (within 6 weeks prior to initial evaluation). This includes all antidepressants and any adjunctive psychotropic medications that are being used to address problems related to mood or anxiety (e.g. antipsychotic medications, mood stabilizers.) This does not include stimulant medications that are being used to treat Attention Deficit Hyperactivity Disorder (ADHD).**
* Current treatment with Bupropion at a dose greater than 150mg per day.
* Current treatment with a stimulant medication as an adjunct medication for depression.***
* Current treatment with a stimulant medication for ADHD above FDA recommended dosages.***

(*) If the participant has an insufficient number of trials in the current episode, then the participant must also have failed ≥1 and ≤4 trials in a previous episode. Subjects who have been unable to complete an antidepressant trial of adequate dose and duration due to intolerance to antidepressant therapy may be included if they have demonstrated intolerance to ≥4 antidepressant medications within one discrete illness episode (current or previous episode as defined above)

(**) If there has been a recent discontinuation of a medication we will require varying lapses of time before study entry depending on medication type as follows: Antidepressant medications = 4 weeks, mood stabilizers (e.g. Lithium, Valproate) = 2 weeks, Antipsychotic medications = 2 weeks, Stimulant medications = 1 week

(***) If participants are being treated with stimulant medications as an adjunct strategy for their depression, we will require them to discontinue the stimulant prior to starting the study treatment and wait 1 week before they begin the study as listed above. If the participant is taking a stimulant medication to treat ADHD, they will be allowed to continue the stimulant medication, as long as the dosage is within FDA recommendations.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Cullen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cullen KR, Jasberg S, Nelson B, Klimes-Dougan B, Lim KO, Croarkin PE. Seizure Induced by Deep Transcranial Magnetic Stimulation in an Adolescent with Depression. J Child Adolesc Psychopharmacol. 2016 Sep;26(7):637-41. doi: 10.1089/cap.2016.0070. Epub 2016 Jul 22. PMID 27447245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Started | 7 | 3 | 14
Completed | 3 | 3 | 8
Not Completed | 4 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT | Total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.07 (1.64) | 17.10 (1.43) | 16.17 (1.52) | 16.3 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 1 | 0 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 2 | 6 | 11
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Child Depression Rating Scale - Revised (CDRS-R)
Description: The Children's Depression Rating Scale-Revised (CDRS-R) is a measure of depression severity in adolescents and children of ages 6 to 12. The measure is completed by a clinician based on interviews with the child/adolescent and their parent. The scale includes 17 symptom areas, each rated on a likert scale ranging from 1 to 5 or 7. Depression severity is indiciated by the CDRS-R raw summary score computed by adding the item responses. The summary score ranges from 17 to 113, with a higher score indicating more severe depression and worse outcome. Change in score for each participant was calculated by subtracting their post-rTMS score from their baseline score, such that a positive value indicates a decrease in score from pre to post-treatment.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 3 | 8
score on a scale | 12.33 (6.03) | 1.33 (3.79) | 22.13 (4.29)

2. Secondary Outcome: Change in Score Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory (BDI-II) is a 21-item self-report measure of depression severity in adolescents and adults. Each item is measured on a likert scale ranging from 0 to 3. A total score is calculated by adding item responses and can range from 0 to 63, with a higher score indicating more severe depression and worse outcome. Change in score for each participant was calculated by subtracting their post-rTMS score from their baseline score, such that a positive value indicates a decrease in score from pre to post-treatment.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 3 | 8
units on a scale | 12.33 (11.02) | 7.33 (5.69) | 10.38 (9.26)

3. Secondary Outcome: Change is Score Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Columbia Suicide Severity Rating Scale (C-SSRS- recent version) is a 10-item measure of suicidal ideation and behavior. Participants were assigned a score between 0 and 8, with higher scores indicating the endorsement of more severe suicidal ideation or behavior (a worse outcome) and a score of "0" indicating no suicidal ideation or behavior (better outcome). Change in score for each participant was calculated by subtracting their post-rTMS score from their baseline score, such that a positive value indicates a decrease in score from pre to post-treatment.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 3 | 8
units on a scale | 4.33 (4.04) | 0.33 (0.58) | 3.38 (3.16)

4. Secondary Outcome: Change in Score Temporal Experience of Pleasure Scale (TEPS)
Description: The Temporal Experience of Pleasure Scale (TEPS) is an 18-item self-report measure of the tendency to anticipate and experience pleasure. Each item is rated on a likert scale ranging from 1 (very false for me) to 6 (very true for me). A total score is calculated by adding item responses and ranges from 18 to 108, such that higher scores indicate greater anticipation and experience of pleasure and better outcome. Change in score for each participant was calculated by subtracting their post-rTMS score from their baseline score, such that a positive value indicates a decrease in score from pre to post-treatment.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 8
units on a scale | -3 (17.06) | 2.5 (21.92) | 0.75 (13.21)

5. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: General Depression
Description: 64-item measure of mood and anxiety disorder symptoms. Each item is rated on a likert scale ranging from 1 (not at all) to 5 (extremely). The measure includes 2 broad subscales of general depresson (20 items; score range: 20-100) and dysphoria (10 items; score range: 10-50) as well as 10 specific symptom scales: Lassitude (6 items; score range: 6-30), Insomnia (6 items; score range: 6-30), Suicidality (6 items; score range: 6-30), Well-Being (8 items; score range: 8-40), Social Anxiety (5 items; score range: 5-25), Appetite Loss (3 items; score range: 3-15), Appetite Gain (3 items; score range: 3-15), Ill Temper (5 items; score range: 5-25), Panic (8 items; score range: 8-40), and Traumatic Intrusions (4 items; score range: 4-20). Subscale scores are calculated by adding responses for items corresponding to the subscale, with higher scores on each subscale except the well-being subscale indicating poorer outcomes. Higher scores on well-being subscale indicates better outcome.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 7.67 (9.29) | 1.5 (16.26) | 17.67 (13.66)

6. Secondary Outcome: Change in Score Young Mania Rating Scale
Description: The Young Mania Rating Scale is a 11-item measure of manic symptoms. Some items are rated on a likert scale ranging from 0 to 4 and some items are rated on a scale ranging from 0 to 8. Total scores range from 0 to 60, with a higher score indiciating higher levels of mania and worse outcome. Change in score for each participant was calculated by subtracting their post-rTMS score from their baseline score, such that a positive value indicates a decrease in score from pre to post-treatment.
Time Frame: Baseline to post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 3 | 7
units on a scale | -0.67 (1.53) | 3 (2.65) | -1.14 (3.08)

7. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Dysphoria
Description: The Inventory of Depression and Anxiety Symptoms (IDAS) is a 64-item measure of mood and anxiety disorder symptoms. Each item is rated on a likert scale ranging from 1 (not at all) to 5 (extremely). The measure includes 2 broad subscales of general depresson (20 items; score range: 20-100) and dysphoria (10 items; score range: 10-50) as well as 10 specific symptom scales: Lassitude (6 items; score range: 6-30), Insomnia (6 items; score range: 6-30), Suicidality (6 items; score range: 6-30), Well-Being (8 items; score range: 8-40), Social Anxiety (5 items; score range: 5-25), Appetite Loss (3 items; score range: 3-15), Appetite Gain (3 items; score range: 3-15), Ill Temper (5 items; score range: 5-25), Panic (8 items; score range: 8-40), and Traumatic Intrusions (4 items; score range: 4-20). Higher scores on each subscale except the well-being subscale indicating poorer outcomes. Higher scores on well-being subscale indicates better outcome.
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 5.67 (6.66) | 5.5 (2.12) | 8.83 (8.61)

8. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Lassitude
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 2.33 (4.16) | 1 (4.24) | 6.67 (4.27)

9. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Insomnia
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 1 (1) | -3.5 (3.54) | 6.33 (6.44)

10. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Suicidality
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 0.67 (2.52) | 2 (0) | 4.17 (4.49)

11. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Appetite Loss
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 0 (0) | -4 (7.07) | 1.33 (5.32)

12. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Appetite Gain
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 1 (1.73) | 0.5 (0.71) | -0.33 (1.97)

13. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Ill Temper
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 0.67 (1.15) | 4.5 (9.19) | 1.17 (3.31)

14. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Well Being
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 2.67 (4.51) | 1 (1.41) | 3.17 (1.72)

15. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Social Anxiety
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 2.67 (4.51) | 1 (1.41) | 3.17 (1.72)

16. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Panic
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 2.67 (0.58) | -0.5 (2.12) | 1.17 (2.14)

17. Secondary Outcome: Change in Score Inventory of Depression and Anxiety Symptoms (IDAS) Subscale: Traumatic Intrusions
Description: as for outcome 7
Time Frame: Baseline to post-rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Period 1: 80% of MT | Period 2: 100% of MT | Period 3: 120% of MT
Number analyzed (Participants) | 3 | 2 | 6
units on a scale | 0.33 (3.51) | 0.5 (0.71) | -1.5 (4.14)

ADVERSE EVENTS:
Time Frame: Baseline to follow-up visit 6, 6 months
Groups:
- Open Label rTMS: All participants who qualify will undergo 6 weeks of open-label rTMS.
  Active Repetitive Transcranial Magnetic Stimulation (rTMS): rTMS applies a pulsatile magnetic field to the scalp which painlessly induces electrical currents to the brain. Typically, rTMS is applied to the dorsolateral prefrontal cortex (DLPFC), a brain region that is hypoactive in depression. Whereas standard rTMS stimulates superficial (1cm depth) cortical areas, recent advances in rTMS coil technology support stimulation of deeper (5 cm depth) limbic structures that are also relevant to depression.
Arm/Group | Open Label rTMS
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label rTMS (N=14)
Suicide ideation (Psychiatric disorders) | 1 (1)
Suicide intent (Psychiatric disorders) | 1 (1)
suicide attempt (Psychiatric disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label rTMS (N=14)
Head and Jaw (General disorders) | 12 (109)
Gastro-intestinal & genito-Urinary (Gastrointestinal disorders) | 3 (14)
Nervous system (Nervous system disorders) | 2 (2)
Psychiatric (Psychiatric disorders) | 7 (19)
skin and subcutaneous tissue (General disorders) | 2 (4)
Cardiovascular (Cardiac disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02611206/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02611206/ICF_000.pdf